CLINICAL TRIAL: NCT02017093
Title: Error Enhancement of the Velocity Component in the Course of Stroke Patients' Reaching Movements - A Pilot Study
Brief Title: Error Enhancement of the Velocity Component
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Tel Aviv University (Other)
Responsible Party: Principal Investigator, Carmeli Eli, Prof, University of Haifa
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UHaifa; CEli (Registry Identifier: Eli Carmeli)
Record Dates: First submitted 2013-06-20; First posted 2013-12-20 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-06

CONDITIONS: Stroke; Hemiparesis
Keywords: CVA, rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Error Enhancement (Experimental): Training of the upper extremity, using a robotic devise with error enhanced forces and traditional therapy.
  Interventions: Device: Error Enhancement
- Control treatment (Experimental): Training of the upper extremity, using a robotic devise without forces applied and traditional therapy.
  Interventions: Device: control treatment

INTERVENTIONS:
Device: Error Enhancement — Patients underwent upper extremity robotic training with the error enhancement effect. Training have focused on hand reaching movements in varity of directions and range of motions.
  Other Names: Experimental: Error Enhancement of the Velocity Component
  Arms: Error Enhancement
Device: control treatment — Patients underwent upper extremity robotic training without the error enhancement effect. Training have focused on hand reaching movements in varity of directions and range of motions.
  Arms: Control treatment

SUMMARY:
The purpose of this pilot study was to explore the impact of enhancement of the velocity component error in the course of reaching movements of the impaired/hemiparetic limb in an acute stroke subject. We hypothesized that the method would shift velocity profiles toward the optimal, resulting in a reduction in error. A prototype robot. This robotic device system has a two-dimensional motor, basic measurement capacities, and a robotic arm which is engaged to the subject's upper-limb in a sitting position.

The enhancement of the velocity component error would shift velocity profiles toward the optimal, resulting in a reduction in error.

DETAILED DESCRIPTION:
The wrist of the subject is connected to the robotic arm by a strip which supports the arm but allows free movements of the wrist. This configuration allows subjects with impaired grasping ability to use the system. A bio-feedback system enables the subject to perform various functional motor tasks that are presented on the screen in front of him. The system's sensors detect motor errors or deviations from an optimal/proper movement trajectory or velocity profile. Any deviation in direction, velocity, acceleration or necessary force from the optimal trajectory results in applied robotic forces that enhance such errors/deviations. The sensors and the applied forces all work and compute in real time, so that the force measurements and the applied force are updated to the executed movement.

ELIGIBILITY:
Inclusion Criteria:

* Single stroke
* Two to three weeks post Stroke
* Able to understand simple commands
* Able to perform some reaching movements with the affected arm.
* No other neurological, neuromuscular, orthopedic disorders and visual deficit

Exclusion Criteria:

* Perceptual, apraxic, or major cognitive deficits,
* Shoulder joint subluxation or pain in the upper-limb, and
* Spasticity > 1 (single muscle Modified Ashworth Scale).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Carmeli, PhD, Principal Investigator — University of Haifa
Locations (1):
- Reuth Medical Center, Tel Aviv, Israel

REFERENCES:
- [Result] Givon-Mayo R, Simons E, Ohry A, Karpin H, Israely S, Carmeli E. A preliminary investigation of error enhancement of the velocity component in stroke patients' reaching movements. International Journal of Therapy and Rehabilitation. 2014;21(4):160-168.
- See also: Click here for more information about this study: http://www.ncbi.nlm.nih.gov/pubmed/18326055 — http://www.ncbi.nlm.nih.gov/pubmed/16249912

RESULTS

PARTICIPANT FLOW:
Groups:
- Error Enhancement: Training of the upper extremity, using a robotic deviset with error enhanced forces and traditional therapy.
  Error Enhancement deXtreme's prototype robot: The subjects were seated on comfortable chairs, individually adjusted, and connected to a manipulandum of deXtreme's prototype robot. We situated the chair so that the computer monitor could be clearly observed by the subject. Each subject's affected extremity was harnessed to a handle connected to a robotic arm accompanying the movement
  Optimal Velocity Profile and Calculation of Error Enhancement: Fugl-Meyer (FM) and the Motor Assessment Scale (MAS) tests were included.
- Control Group: Traditional Therapy: Training of the upper extremity, using a robotic deviset without forces applied and traditional therapy.
  Error Enhancement deXtreme's prototype robot: The subjects were seated on comfortable chairs, individually adjusted, and connected to a manipulandum of deXtreme's prototype robot. We situated the chair so that the computer monitor could be clearly observed by the subject. Each subject's affected extremity was harnessed to a handle connected to a robotic arm accompanying the movement
  Optimal Velocity Profile and Calculation of Error Enhancement: Fugl-Meyer (FM) and the Motor Assessment Scale (MAS) tests were included.
Period: Overall Study
Arm/Group | Error Enhancement | Control Group: Traditional Therapy
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study; Control: Patients admitted to rehabilitation center after a stroke.
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.9) | 57.33 (7.3) | 59.14 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 3 | 6
Fugl-Meyer assessment score [Mean (Standard Deviation); unit: units on a scale] | 53.2 (3.26) | 54.3 (5.43) | 53.7 (4.36)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Average Movement Trajectory Error From T1 to T2
Description: While reaching, people have typical movement pattern of trajectory, moving the end-effector (hand) in straight line. The abnormal motor control after a stroke may cause these patients to deviate from this pattern. Our robotic device enabled us to measure the magnitude of the deviation from the optimal profile of healthy people. This was followed by a calculation of the average error the paricipants made in each treatment session. So we finally recieved a score of the average magnitude of trajectory error the participants made through a treatment session. Each treatment seesoin composed of about 100 reaching movements. The outcome measure expresses the change in the movement error from T1 to T2.
Time Frame: The outcome was assessed at the begining of the rehabilitation (T1) and about 5 weeks later at the end of rehabilitation (T2).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Error Enhancement | Control Group: Traditional Therapy
Number analyzed (Participants) | 4 | 3
cm | 2.31 (1.52) | 2.4 (1.2)

2. Primary Outcome: Fugl-Meyer Assessment Score
Description: The Fugl-Meyer assessment score (FM) is a zero (disabaled function) to 66 points (high level of function) scale that evaluates the level of the motor impairment of the upper extremity, in stroke patients.
Time Frame: The measured assessed at the begining of the rehabilitation (T1) and about 5 weeks later at the end of the rehabilitation (T2).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group: Training of the upper extremity, using a robotic devise without forces applied and traditional therapy.
  control treatment: Patients underwent upper extremity robotic training without the error enhancement effect. Training have focused on hand reaching movements in varity of directions and range of motions.
Arm/Group | Error Enhancement | Control Group
Number analyzed (Participants) | 4 | 3
units on a scale
  Fugl-Meyer score at T1 | 53.2 (3.26) | 54.33 (5.43)
  Fugl-Meyer score at T2 | 56.75 (2.38) | 55.33 (4.49)

ADVERSE EVENTS:
Time Frame: There were no adverse events during the whole trial.
Description: Adverse events for all the study participants, were monitored seperately for each of the participants, at the end of the last treatment session.
  At the end of the study no adveres events were reported from any of investigators to the ethics committee of the rehabilitation institute.
Arm/Group | Error Enhancement | Control Group: Traditional Therapy
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No